CLINICAL TRIAL: NCT01738854
Title: The Comparison of Airway Sealing With the Laryngeal Mask Airway (LMA) Supreme at Different Intracuff Pressure in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1-2012-0043
Record Dates: First submitted 2012-11-22; First posted 2012-11-30 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: General Anesthesia
Keywords: laryngeal mask airway supreme; airway sealing; intracuff pressure

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- intra-cuff pressure 40 cmH2O (Experimental)
  Interventions: Procedure: intracuff pressure by cuff pressure manometer
- intra-cuff pressure 60 cmH2O (Active Comparator)
  Interventions: Procedure: intracuff pressure by cuff pressure manometer
- intra-cuff pressure 80 cmH2O (Active Comparator)
  Interventions: Procedure: intracuff pressure by cuff pressure manometer

INTERVENTIONS:
Procedure: intracuff pressure by cuff pressure manometer — 36 patients are randomly allocated according to random sequence of the intracuff pressure 40, 60 and 80 cmH2O. After insertion of LMA supreme, we confirm adequate ventilation. And then we measure OLP and leakage volume at intra-cuff pressure 40, 60 and 80 cmH2O adjusted by cuff pressure manometer according to random sequence of the intracuff pressure.

SUMMARY:
The laryngeal mask airway (LMA) supreme is a relatively new single-use supraglottic airway with modification. The parameters about airway sealing such as oropharyngeal leak pressure (OLP) and leakage volume are important markers of efficacy and safety when using the supraglottic airway. The airway sealing is related to the intracuff pressure of laryngeal mask airway. The aim of this study is to compare the airway sealing of the LMA supreme at various intracuff pressure in children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (less than 108months of age)
* scheduled for elective surgery undergoing general anesthesia using LMA supreme 1.5-2.5

Exclusion Criteria:

* Patients with an abnormal airway,
* reactive airway disease,
* gastroesophageal reflux disease,
* chronic respiratory disease,
* a history of an upper respiratory tract infection

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The oropharyngeal leak pressure volume | approximately 5 minutes after adjusting intracuff pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Zhang L, Seet E, Mehta V, Subramanyam R, Ankichetty SP, Wong DT, Chung F. Oropharyngeal leak pressure with the laryngeal mask airway Supreme at different intracuff pressures: a randomized controlled trial. Can J Anaesth. 2011 Jul;58(7):624-629. doi: 10.1007/s12630-011-9514-6. Epub 2011 Apr 30. PMID 21533663